CLINICAL TRIAL: NCT06450353
Title: Prospective Evaluation of Disparities in Provision of Allogeneic Transplantation
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0253; NCI-2024-04790 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-31; First posted 2024-06-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Allogeneic Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective evaluation: Participants are expected to be in this research study for up to 2 years after the participants bone marrow transplantation. However, your active participation will only last 1 day, when you sign the consent form and complete a questionnaire about your demographic information and ancestry (family ethnicity). For the rest of the study, information about the participants medical history, choice of bone marrow donor, and health outcomes will be collected from your medical record.
  Interventions: Behavioral: Patient Ancestry Questionnaires

INTERVENTIONS:
Behavioral: Patient Ancestry Questionnaires — Participants will be asked to complete a demographics and ancestry questionnaire at the baseline visit before you and your doctor select bone marrow donation candidates.

SUMMARY:
To look at the effect of a recipient's ancestry and socio-economic status on their choice of bone marrow transplantation donor cells and their chance of receiving genetically similar (allogeneic) bone marrow cells versus cells that are not genetically similar (allograft).

DETAILED DESCRIPTION:
Primary Objectives To prospectively evaluate graft options and choice of donor by patient ancestry and SES for allograft candidates at MDACC.

Secondary Objectives

* To prospectively evaluate time to transplant for allograft candidates at MDACC.
* To evaluate treatment-related mortality for allograft candidates at MDACC.
* To assess overall survival for allograft candidates at MDACC.
* To prospectively evaluate receipt of preferred unrelated donor for allograft recipients at MDACC.
* To evaluate receipt of an optimal graft for allograft recipients at MDACC.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Candidate for allogeneic transplantation

Exclusion Criteria:

1) Allogeneic stem cell transplantation not medically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Ancestry Questionnaire | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Fingrut, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org